CLINICAL TRIAL: NCT03859440
Title: Three-month Clinical Evaluation of DSiHy Daily Disposable Silicone Hydrogel Contact Lenses
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: HOYA Lamphun Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: HOYA-3601
Record Dates: First submitted 2019-02-20; First posted 2019-03-01 (Actual); Last update posted 2019-03-07 (Actual); Status verified 2019-03

CONDITIONS: Contact Lenses

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DSiHy (test lens) (Experimental)
  Interventions: Device: DSiHy Silicone hydrogel soft contact lens
- Silicone hydrogel soft contact lens CE-marked for daily use (Active Comparator)
  Interventions: Device: CE-marked Silicone hydrogel soft contact lens

INTERVENTIONS:
Device: DSiHy Silicone hydrogel soft contact lens — •Device: DSiHy (test lens) Silicone hydrogel soft contact lens for daily disposable wear.
  Arms: DSiHy (test lens)
Device: CE-marked Silicone hydrogel soft contact lens — ・Device: Silicone hydrogel soft contact lens CE-marked for daily disposable wear.
  Other Name : MyDay
  Arms: Silicone hydrogel soft contact lens CE-marked for daily use

SUMMARY:
The purpose of this study is to evaluate the clinical performance of two daily disposable silicone hydrogel contact lenses. One of these lenses, the 'test' lens is an investigational product. This means that it has not yet been approved for commercial use and is not available for sale. The other lens (control) is a commercially available contact lens.

The results of this study will be analysed to determine how the 'test' lens compares with the 'control' lens. The control lens has been chosen because it is a market leader and is well tried and tested.

Participants who are in this study will need to have healthy eyes, except for the need to correct their eyesight. Up to 90 people who are aged 20 years or older will be considered for participation in this study. The study is designed to be approximately 3 months long.

ELIGIBILITY:
Inclusion Criteria:

* Be aged 20 years or more.
* Sign written informed consent.
* Be a currently adapted soft contact lens wearer (i.e. be wearing lenses at least 1 month prior to enrolment).
* Contact lens sphere requirement between -1.00 to -6.00 D (inclusive).
* Refractive astigmatism (if present) less than or equal to 0.75 D in both eyes.
* Be correctable by sphero-cylindrical refraction to 6/7.5 (+0.10 logMAR 0.8 decimal) or better in each eye.
* Require visual correction in both eyes (monovision allowed, no monofit.

Exclusion Criteria:

* Require toric or multifocal contact lenses.
* Concurrent ocular medication.
* Using systemic or topical medications that will in the investigator's opinion affect ocular physiology or contact lens performance.
* Any systemic illness affecting contact lens wear or the medical treatment of which would affect vision or successful lens wear (including diabetes).
* Clinically significant (≥Grade 2) corneal staining, corneal edema, corneal vascularization, tarsal abnormalities, bulbar hyperemia, limbal hyperemia, or any other abnormality of the cornea that would contraindicate contact lens wear.
* History of herpetic keratitis.
* Pathological dry eye.
* Aphakia or amblyopia.
* History of refractive surgery, keratoconus or other corneal irregularity.
* Pregnancy, lactating or planning a pregnancy at the time of enrolment.
* Participation in any concurrent clinical trial or within the last 30 days.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2019-05 (Estimated); Primary Completion 2019-10 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
Lens-related ocular adverse events requiring temporary or permanent discontinuation (resting eyes) as a proportion of follow-up eye examinations. | 13 week visit
Proportion of eyes with visual acuity corrected to 6/6 or better (1.0 decimal) at each visit. | 13 week visit
Proportion of eyes with best sphere-corrected visual acuity of 6/6 or better (1.0 decimal) at each visit. | 13 week visit

SECONDARY OUTCOMES:
The following variables will be compared between lens types: Corneal staining - type (mean grade, 0-4) | 13 week visit
  Assessed by sector with fluorescein, blue light, yellow filter and full beam using medium magnification.
  0 NONE: No staining
  1. Micropunctate - Punctate staining, minor localized or scattered in on one or two quadrants
  2. Macropunctate - Coalescent punctate staining, localized in one or two quadrants
  3. Widespread coalescent punctate staining in more than two quadrants
  4. Confluent staining or erosion (usually accompanied by hyperemia)
The following variables will be compared between lens types: Limbal hyperemia (grade, 0-4) | 13 week visit
  Assessed using slit lamp with white light, low-medium magnification 0 NONE: No injection present
  1. TRACE: Slight limbal (mild segmented), bulbar (mild regional), and/or palpebral injection
  2. MILD: Mild limbal (mild circumcorneal), bulbar (mild diffuse) injection
  3. MODERATE: Significant limbal (marked segmented), bulbar (marked regional or diffuse) injection
  4. SEVERE: Severe limbal (marked circumcorneal), bulbar (diffuse episcleral or scleral) injection
The following variables will be compared between lens types: Bulbar hyperemia (grade, 0-4). | 13 week visit
  Assessed using slit lamp with white light, low-medium magnification 0 NONE: No injection present
  1. TRACE: Slight limbal (mild segmented), bulbar (mild regional), and/or palpebral injection
  2. MILD: Mild limbal (mild circumcorneal), bulbar (mild diffuse) injection
  3. MODERATE: Significant limbal (marked segmented), bulbar (marked regional or diffuse) injection
  4. SEVERE: Severe limbal (marked circumcorneal), bulbar (diffuse episcleral or scleral) injection
The following variables will be compared between lens types: Comfort (0-10) | 13 week visit
  Assessed by subject. 0 to 10 scale 10 = cannot be felt 0 = painful
The following variables will be compared between lens types: Visual acuity (logMAR VA) | 13 week visit
The following variables will be compared between lens types: Wettability (0-4). | 13 week visit
  Lens surface wettability rated on the appearance of the lens surface and the drying time viewed with a slit lamp under low magnification.
  0 VERY POOR: Immediately displaying non-wetting areas on lens surface.
  1. POOR: Irregular surface appearance; drying time <interblink period.
  2. ACCEPTABLE: Smooth surface appearance immediately after the blink becoming irregular with time; drying time >interblink period.
  3. GOOD: Typical lens appearance with long drying time.
  4. EXCELLENT: Appearance of a healthy cornea with very long drying time.

CONTACTS AND LOCATIONS:
Overall Officials: Graeme Young, Dr, Principal Investigator — Visioncare Research Ltd.

IPD SHARING:
Plan to Share IPD: No